CLINICAL TRIAL: NCT07107815
Title: A Study On The Prediction of Neoadjuvant Efficacy And Heterogeneity For Rectal Cancer Based On MR Cytometry Imaging and Deep-radiomics
Brief Title: A Study On The Prediction of Neoadjuvant Efficacy For Rectal Cancer Based On MR Cytometry Imaging and Deep-radiomics
Status: Enrolling by invitation | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: NCC2025C-250
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer, Adenocarcinoma
Keywords: rectal cancer; MR cytometry imaging; deep-radiomics; neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study employed MR cytometry imaging combined with deep-radiomic research methods to predict the heterogeneity of rectal cancer, and constructed a model to predict the sensitivity to neoadjuvant therapy and potential mechanisms, assisting clinicians in early identification of high-risk tumors and patients with treatment-susceptible rectal cancer, and selecting individualized treatment plans, thereby improving patient prognosis. To this end, the investigators need to collect the clinical diagnosis and treatment data of patients, surgical and biopsy pathological information, pre-treatment rectal MRI images and colonoscopy biopsy tissue sections, and follow up on the surgical pathological results and recurrence of patients. This study is a non-interventional diagnostic study, which does not interfere with the routine diagnosis and treatment of patients, does not affect any medical rights of patients, and does not increase any medical risks.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed rectal adenocarcinoma without previous treatment
* Complete radical surgery in the institute
* Complete rectal MRI within 2 weeks before surgery

Exclusion Criteria:

* Concomitant malignancies or systemic disease
* Inadequate MR image quality for analysis
* Incomplete clinicopathological data
* Loss of follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese patients diagnosed with rectal cancer through pathological examination
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | One month after surgery
Pathological tumor regression grade | One month after surgery
progression-free survival | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months

SECONDARY OUTCOMES:
Pathological differentiation grade | One month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhao Q, Shi D, Zhong H, Jin C, Wang Z, Shi Z, Li L, Wang B, Jiang Y, Feiweier T, Xu J, Guo H, Zhang H. The predictive value of MR cytometry in histological differentiation of rectal cancer: an exploratory study. Eur Radiol. 2026 Jan 30. doi: 10.1007/s00330-026-12341-w. Online ahead of print. PMID 41617831